CLINICAL TRIAL: NCT03676829
Title: Embolization for the Treatment of Pain Secondary to Adhesive Capsulitis
Acronym: AES
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vascular Institute of Virginia (Other)
Collaborators: Terumo Medical Corporation (Industry)
Responsible Party: Principal Investigator, Sandeep Bagla, Principal Investigator, Sandeep Bagla, MD, Vascular Institute of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G180115; 20181853 (Other: WIRB)
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Frozen Shoulder; Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Arterial Embolization of the Shoulder (AES) (Experimental): Patients in this study will receive the arterial embolization of the shoulder (AES) procedure. The primary aims will be to determine if arterial embolization of the shoulder (AES) will reduce pain and improve range of motion (ROM) caused by adhesive capsulitis.
  Interventions: Device: Arterial Embolization of the Shoulder

INTERVENTIONS:
Device: Arterial Embolization of the Shoulder — Arterial Embolization of the Shoulder (AES) is a new procedure that is being used to reduce pain and improve range of motion (ROM) caused by adhesive capsulitis. Embolization is a procedure where physicians intentionally block the blood vessels to specific areas of the body to prevent blood flow to that region. By doing this, the decrease in blood flow will decrease the size of the area of interest. In this case, the goal is to decrease the size of inflammatory tissue around the shoulder, resulting in improvement of pain, stiffness and from adhesive capsulitis.

SUMMARY:
This study is to test a new treatment method, arterial embolization of the shoulder (AES), to reduce the severity of pain and improve range of motion (ROM), and to see if it can be performed safely.

DETAILED DESCRIPTION:
Purpose: The primary aims of this study are to determine if arterial embolization of the shoulder will reduce the severity of pain as well improve Range of Motion (ROM) caused by adhesive capsulitis and if it can be performed safely. The secondary aim is to determine if AES can result in the decreased necessity for ongoing conservative therapies, such as medication therapy and joint injections.

Participants: Twenty patients with adhesive capsulitis, resulting in shoulder pain that is refractory to conservative therapies, who are not planning to undergo surgery within 6 months.

Procedures (methods): This will be an open label 24-month pilot study with a small population undergoing AES to determine safety and efficacy. Clinical procedures and evaluations will consist of a preoperative screening assessment to determine if the potential study subject meets the inclusion and exclusion criteria, enrollment, surgical procedure for arterial embolization of the shoulder, and follow-up visits at 24 hours, 1, 3 & 6 months. An MRI will be performed at the 1-month visit to detect a change in capsular vascularity and to exclude complication.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe shoulder pain (VAS greater than 40mm), and
* diagnosis of adhesive capsulitis, and
* age > 21, and
* pain refractory to at least 30 days of conservative therapy (pain medications, physical therapy, etc.)

Exclusion Criteria:

* current local infection, or
* life expectancy less than 6 months, or
* known advanced atherosclerosis, or
* rheumatoid or infectious arthritis, or
* prior shoulder replacement surgery, or
* uncorrectable coagulopathy as defined by INR > 2.5 or platelets < 30,000, or
* iodine allergy resulting in anaphylaxis, or
* renal dysfunction as defined by GRF of < 45, or
* contraindication for magnetic resonance imaging, or
* known complete full thickness tear of rotator cuff, or
* currently pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient Pain | 6 months
  The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain". Pain will be assessed at each of the patient's follow-up visits and used to measure the change from baseline (prior to the AES procedure). The investigators will use this to measure if the patient's pain level decreases.
Patient Function | 6 months
  The American Shoulder and Elbow Surgeons Shoulder Score (ASES) will be used to measure function. This is a score derived from a questionnaire in which the patient answers questions regarding range of motion, stiffness, and pain and how it affects the ability to function.

SECONDARY OUTCOMES:
Reduction in Medication | 6 months
  Reduction in the number or strength of previously initiated medical therapy (e.g. NSAIDs).
Improvement of Range of Motion | 6 months
  Patients' range of motion will be assessed prior to undergoing embolization and at 1,3, and 6 month follow ups.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Bagla, MD, Principal Investigator — Vascular Institute of Virginia
Locations (1):
- Vascular Institute of Virginia, Woodbridge, Virginia, United States

IPD SHARING:
Plan to Share IPD: No